CLINICAL TRIAL: NCT05617573
Title: Correlations Between Microscopic Features of Synovium and Clinical Parameters in Patients With Advanced Osteoarthritis
Brief Title: Synovitis in Patients With Osteoarthritis
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Xiang Shuai, MD, Principal Investigator, The Affiliated Hospital of Qingdao University
Other Study IDs: OASynoviumAHQD
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergone TKA due to advanced knee osteoarthritis
  Interventions: Procedure: Total knee arthroplasty due to advanced osteoarthritis.

INTERVENTIONS:
Procedure: Total knee arthroplasty due to advanced osteoarthritis. — Postoperative usage of intravenous methylprednisolone

SUMMARY:
To study synovial membrane (SM) inflammation in suprapatellar fossa in advanced knee osteoarthritis (OA), and to correlate the pathological features with clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective, unilateral, primary TKA for advanced osteoarthritis.

Exclusion Criteria:

- revisions, bilateral procedures, alcohol or medical abuse, administration of any glucocorticoids during the 3 months prior to surgery, and/or a history of serious cardiac or cerebrovascular problems, severe liver or kidney failure, and/or connective tissue disease including rheumatoid arthritis, ankylosing spondylitis, and systemic lupus erythematosus.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between pathological features and clinical scores | 1 day.
Correlation between pathological features and laboratory index | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No